CLINICAL TRIAL: NCT04738435
Title: Safety of the Sputnik V Vaccine in Health Personnel of Private Effectors of the City of Buenos Aires, Argentina
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government)
Responsible Party: Principal Investigator, VANINA LAURA PAGOTTO, Vanina Pagotto, Hospital Italiano de Buenos Aires
Other Study IDs: 3876
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: Population Surveillance; COVID-19 Vaccines; adverse effects
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main of the study is to describe the incidence in health personnel who present events supposedly attributed to vaccines and immunizations after having received the two components of the Sputnik V vaccine, with the information obtained thanks to the participation of health workers in actively reporting their health status.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends vaccination against coronavirus disease 19 (COVID-19) as a fundamental primary prevention tool to limit the health and economic effects of the pandemic. having effective and safe vaccines in the short term,will help to reduce the incidence of illness, hospitalizations and deaths related to COVID-19 and help to gradually restore a new normality in the functioning of our country.

On December 23, within the framework of Law 27573, the National Administration of Medicines, Food and Medical Technology submitted the report on the Sputnik V vaccine to the Ministry of Health of the Nation to advance in the Emergency Authorization.

The National Government ensures the processes to reach the standards of safety and efficacy for the entire Argentine territory, being vaccination in stages, free, voluntary and independent of the history of having suffered the disease.

For the surveillance of vaccine safety, the Strategic Plan proposes to health effectors "To develop a specific plan for intensified passive and active surveillance of vaccine safety, which allows the continuous analysis of the notifications of Events Supposedly Attributed to Vaccines and Immunizations.

The Ministry of Health of Buenos Aires City articulated the public and private effectors for the epidemiological follow-up of the personnel vaccinated with the first vaccines in relation to the frequency of Events Supposedly Attributed to Vaccines and Immunizations.

The main of the study is to describe the incidence in health personnel who present events supposedly attributed to vaccines and immunizations after having received the two components of the Sputnik V vaccine, with the information obtained thanks to the participation of health workers in actively reporting their health status.

ELIGIBILITY:
Inclusion Criteria:

* health workers who agree to receive the sputnik V vaccine

Exclusion Criteria:

* health workers who have a contraindication to receive the sputnik V vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: health workers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of events supposedly attributed to vaccines and immunizations after Sputnik V | From first doses up to 10 days
  Incidence of events supposedly attributed to vaccines and immunizations after the fist and second doses of Sputnik V in in health personnel

CONTACTS AND LOCATIONS:
Overall Officials: Vanina pagotto, Msc, Principal Investigator — Hospital Italiano de Buenos Aires; Silvana Figar, Msc, Study Chair — Hospital Italiano de Buenos Aires; Mercedes Soriano, Study Chair — Hospital Italiano de Buenos Aires; Analia Ferloni, MD, Study Chair — Hospital Italiano de Buenos Aires; Valeria Aliperti, Msc, Study Chair — Hospital Italiano de Buenos Aires; Morena Diaz, Study Chair — Hospital Italiano de Buenos Aires; Nahuel Braguisnky, Study Chair — Hospital Italiano de Buenos Aires; Maria Isabel González, Study Chair — Hospital Italiano de Buenos Aires; Maria Ines Staneloni, MD, Study Chair — Hospital Italiano de Buenos Aires; Valeria Asprea, MD, Study Chair — Hospital Italiano de Buenos Aires; Paula Zingoni, MD, Study Chair — Ministry of Health of the Government of the City of Buenos Aires; Hernan Michelangelo, MD, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Result] Di Pasquale A, Bonanni P, Garcon N, Stanberry LR, El-Hodhod M, Tavares Da Silva F. Vaccine safety evaluation: Practical aspects in assessing benefits and risks. Vaccine. 2016 Dec 20;34(52):6672-6680. doi: 10.1016/j.vaccine.2016.10.039. Epub 2016 Nov 8. PMID 27836435
- [Result] Herve C, Laupeze B, Del Giudice G, Didierlaurent AM, Tavares Da Silva F. The how's and what's of vaccine reactogenicity. NPJ Vaccines. 2019 Sep 24;4:39. doi: 10.1038/s41541-019-0132-6. eCollection 2019. PMID 31583123
- [Result] Virtanen M, Peltola H, Paunio M, Heinonen OP. Day-to-day reactogenicity and the healthy vaccinee effect of measles-mumps-rubella vaccination. Pediatrics. 2000 Nov;106(5):E62. doi: 10.1542/peds.106.5.e62. PMID 11061799
- [Result] Mitchell TC, Casella CR. No pain no gain? Adjuvant effects of alum and monophosphoryl lipid A in pertussis and HPV vaccines. Curr Opin Immunol. 2017 Aug;47:17-25. doi: 10.1016/j.coi.2017.06.009. Epub 2017 Jul 17. PMID 28728074
- [Result] Sadoff J, Le Gars M, Shukarev G, Heerwegh D, Truyers C, de Groot AM, Stoop J, Tete S, Van Damme W, Leroux-Roels I, Berghmans PJ, Kimmel M, Van Damme P, de Hoon J, Smith W, Stephenson KE, De Rosa SC, Cohen KW, McElrath MJ, Cormier E, Scheper G, Barouch DH, Hendriks J, Struyf F, Douoguih M, Van Hoof J, Schuitemaker H. Interim Results of a Phase 1-2a Trial of Ad26.COV2.S Covid-19 Vaccine. N Engl J Med. 2021 May 13;384(19):1824-1835. doi: 10.1056/NEJMoa2034201. Epub 2021 Jan 13. PMID 33440088
- [Result] Jackson LA, Anderson EJ, Rouphael NG, Roberts PC, Makhene M, Coler RN, McCullough MP, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott A, Flach B, Doria-Rose NA, Corbett KS, Morabito KM, O'Dell S, Schmidt SD, Swanson PA 2nd, Padilla M, Mascola JR, Neuzil KM, Bennett H, Sun W, Peters E, Makowski M, Albert J, Cross K, Buchanan W, Pikaart-Tautges R, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020 Nov 12;383(20):1920-1931. doi: 10.1056/NEJMoa2022483. Epub 2020 Jul 14. PMID 32663912
- [Result] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- See also: World Health Organization — https://www.who.int/
- See also: Technical report on the regulatory profile on authorization for the use of Sputnik V vaccine within the framework of the Law 27.573 National Administration of Drugs, Food and Medical Technology. Argentina — https://www.argentina.gob.ar/noticias/informe-de-la-anmat-sobre-la-vacuna-sputnik-v
- See also: Argentine Ministry of Health — https://www.argentina.gob.ar/salud
- See also: Strategic Plan for vaccination against COVID-19 in Argentina — https://www.argentina.gob.ar/coronavirus/vacunacion
- See also: Online help Integrated Argentine Health Information System — https://sisa.msal.gov.ar/sisadoc/docs/050203/nomivac_home.jsp
- See also: Argentine citizen digital profile to manage procedures and receive personalized information — https://www.argentina.gob.ar/miargentina
- See also: Epidemiological approach to risk in health care. University of San Carlos of Guatemala. Faculty of Medical Sciences — https://saludpublicayepi.files.wordpress.com/2012/08/enfoque.pdf
- See also: National Administration of Drugs, Food and Medical Technology. Argentina — https://www.argentina.gob.ar/anmat